CLINICAL TRIAL: NCT04226352
Title: An Open-Label Tolerance Study of Three Dosing Regimens of Dextromethorphan (DXM) Reportedly Used in Major Depressive Disorder
Brief Title: Three Dosing Regimens of Dextromethorphan (DXM) Reportedly Used in Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00192193
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-01

CONDITIONS: MDD; Treatment Resistant Depression; Smoking Cessation; Smoking
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Smoking Cessation; Smoking | interventions — Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dose 1 (Experimental): 60 mg DXM a day for 28 days
  Interventions: Drug: Dextromethorphan
- Dose 2 (Experimental): 300 mg DXM every 2 weeks for 28 days.
  Interventions: Drug: Dextromethorphan
- Dose 3 (Experimental): 300mg DXM once, with 60mg DXM daily afterwards
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — Dextromethorphan will be administered and its tolerability evaluated.

SUMMARY:
This is an open-label dosing pilot study of 15 patients aged 18-50 years of age with diagnoses of Major Depressive Disorder (MDD) randomized to 1 of 3 treatment arms.

The study will consist of a screening evaluation performed within the course of 2 weeks, followed by an active treatment period of 28 days where treatment arm 1 will take a supervised dose of 300mg DXM every 14 days for 28 days, treatment arm 2 will take the FDA approved maximum daily ingestion for cough (60mg DXM) daily for 28 days, and treatment arm 3 will take 1 supervised dose of 300mg DXM and 60mg for the remaining 28 days. After the active treatment period, subjects will be followed for 65 days with safety and psychiatric assessments at designated timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a man or woman, 18 to 50 years, inclusive
* Subject must meet Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-V) criteria for MDD without psychotic features based on clinician assessment.
* Subjects must have undergone 3 or fewer antidepressant trials
* Subjects must have moderate to severe depression as determined by a screening Montgomery-Åsberg Depression Rating Scale (MADRS) score of 20 or greater

Exclusion Criteria:

* Subject has a current diagnosis of Bipolar Affective Spectrum Disorder, obsessive compulsive disorder, or a DSM-V personality disorder
* Subject has had an incomplete response to more than 3 antidepressant trials
* Subject cannot tolerate 60mg DXM as determined by study physician
* Subject meets DSM-5 severity criteria for moderate or severe substance or alcohol use disorder within 6 months of screening, excluding caffeine or nicotine
* Subject has a current clinical diagnosis of autism, dementia, or intellectual disability
* Subject has history of psychosis not attributable to organic/metabolic causes
* Subject has a history of serotonin syndrome or sensitivity
* Subject has taken venlafaxine or a monoamine oxidase inhibitor (MAOI) within 4 weeks prior to screening
* Subject is actively taking an opiate antagonist for any indication
* Subject is taking a higher-than-recommended dosage of serotonergic antidepressant [including but not limited to selective serotonin reuptake inhibitor (SSRI), serotonin-norepinephrine reuptake inhibitor (SNRI), serotonin partial agonist/reuptake inhibitor (SPARI), serotonin antagonist and reuptake inhibitor (SARI) within 4 weeks prior to screening
* Subject is actively suicidal
* Subject has participated in another clinical drug trial within 6 months prior to screening
* Subject has a history or current signs of liver or renal insufficiency
* Subject has a clinically significant condition of any organ system that might adversely impact subject health upon consumption of DXM
* Subject has previous history of intolerance to ketamine or its enantiomers
* Subject has previous history of incomplete antidepressant response to ketamine or its enantiomers
* Subject is currently using DXM for any indication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Time to All-Cause Discontinuation of Dextromethorphan | Up to 90 days
  This will be measured in days from the first administration of the drug until discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Kumar, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Department of Psychiatry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No